CLINICAL TRIAL: NCT00652457
Title: A Pilot Study of Memantine for Cognitive and Behavioral Dysfunction in Huntington's Disease"
Brief Title: Study of Memantine to Treat Huntington's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jody Corey-Bloom, MD, PhD (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Jody Corey-Bloom, MD, PhD, Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEM-HD
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine (Experimental): Memantine 10 mg BID for three months
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): Placebo 10 mg BID for three months
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — 10 mg BID x 3 months
  Other Names: Namenda

SUMMARY:
To determine if memantine in doses of 10 mg BID affects memory, cognition, and behavior in patients with Huntington's disease (HD).

DETAILED DESCRIPTION:
Results of several published clinical trials suggest that memantine has a beneficial effect in dementing conditions, such as Alzheimer's disease; however, the effects of memantine on cognitive and behavioral function in HD are unknown. Our hypotheses are that HD patients who are administered memantine will show improved performance on psychometric tests of memory and executive functions in addition to behavior and that patients treated with memantine will show more improvement after six months than after three months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 or older.
* Diagnosis of HD with current complaints of memory or concentration difficulties.
* Dementia Rating Scale score of <129, to ensure that patients have sufficient cognitive impairment.
* Adequate visual and auditory acuity to allow neuropsychological testing.
* Good general health with no additional diseases expected to interfere with the study.
* Patient is not institutionalized.
* Sufficient English skills to complete all testing without assistance of an English language interpreter.
* Availability of a responsible caregiver who agrees to supervise administration of study drug, monitor the patient's compliance and adverse events, and accompany the patient to all clinic visits.

Exclusion Criteria:

* 1. Any significant neurologic disease other than HD.
* Severe psychotic features or other severe psychiatric problems within the last three months which could lead to difficulty complying with the protocol.
* History of alcohol or substance abuse within the past two years (DSM IV criteria).
* Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol.
* History of MI in the past year or head trauma with loss of consciousness greater than 20 minutes.
* Insulin-requiring diabetes.
* Use of any FDA approved cognitive enhancing prescription medications or investigational drugs within 30 days.
* Use of ginkgo biloba or DHEA within four weeks prior to baseline.
* Use of narcotic analgesics within 4 weeks prior to baseline.
* Patients who, in the investigator's opinion, would not comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-11-23 (Actual); Primary Completion 2009-10-28 (Actual); Study Completion 2009-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California, San Diego, La Jolla, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Hospital, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-five participants were screened for eligibility; 6 individuals failed screening by not meeting inclusion criteria forthe study; 9 declined to participate. Fifty participants were then randomized.
Groups:
- Memantine, Then Memantine: Participants first received 10 mg Memantine twice a day for 3 months. No washout. Participants continued on 10 mg Memantine twice a day for another 3 months.
- Placebo, Then Memantine: Participants first received Placebo twice a day for 3 months. No washout. Participants then received 10 mg Memantine twice a day for 3 months.
Period: Overall Study
Arm/Group | Memantine, Then Memantine | Placebo, Then Memantine
Started | 23 | 27
Completed | 23 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Total of all reporting groups due to age of study. Data was not analyzed per arm.
Arm/Group | All Participants
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (NA) — Due to the age of this study (2003), the only age-related results available is the mean age of all participants. The standard deviation was not calculated and the data is no longer accessible.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in the Hopkins Verbal Learning Test - Revised for Delayed Recall (HVLT-R-delayed Recall)
Description: The HVLT-R consists of 3 parts. Free recall has a range of 0 to 36, delayed recall has a range from 0 to 12, and delayed recognition has a range of -12 to 12. Higher scores indicating better function in all 3 parts. Standardized scores are used by calculating an average standardized z score for each part of the HVLT-R. Change is calculated by subtracting baseline value from the respective later time point value. Imputation methods were used to determine values for all alive patients missing the post-baseline assessments. This tool is being used to measure cognitive function, specifically memory.
Time Frame: Baseline, 3 months from start of drug treatment, 6 months from start of drug treatment
Population: Due to the age of this study (2003), the data is no longer accessible. We have been moved a number of times in 17 years and that data has been lost.
Arm/Group | Memantine, Then Memantine | Placebo, Then Memantine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Neuropsychiatric Inventory (NPI)
Description: The Neuropsychiatric Inventory (NPI) assesses the frequency and severity of 12 common behavioral symptoms in dementia.
  The NPI Score is calculated by multiplying the total reported frequency by the severity score, with a theoretical range of 0-1704: high scores indicating greater frequency by severity.
  The change between 2 or more time points is being reported.
Time Frame: Baseline, 3 months from start of drug treatment, 6 months from start of drug treatment
Population: as for outcome 1
Arm/Group | Memantine, Then Memantine | Placebo, Then Memantine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Due to the age of this study (2003), the data regarding individual arms is no longer accessible. We have been moved a number of times in 17 years and that data has been lost.
Arm/Group | Memantine, Then Memantine | Placebo, Then Memantine
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/27
Other Adverse Events (participants affected / at risk) | 4/23 | 1/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine, Then Memantine (N=23) | Placebo, Then Memantine (N=27)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the age of this study (2003), the data is no longer accessible. We have been moved a number of times in 17 years and that data has been lost. The only information we have was provided here in the Results section.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes